CLINICAL TRIAL: NCT00723931
Title: PegIntron Injection Surveillance Plan
Brief Title: PegIntron Injection Surveillance Plan (Study P04123)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P04123
Record Dates: First submitted 2008-07-25; First posted 2008-07-29 (Estimated); Results first posted 2010-12-13 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-11

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2b

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants with Chronic Hepatitis C: Surveillance will be conducted at digestive departments of internal medicine in university or general hospitals where participants with Chronic Hepatitis C are generally treated.
  Interventions: Biological: Peginterferon alfa-2b (SCH 54031)

INTERVENTIONS:
Biological: Peginterferon alfa-2b (SCH 54031) — Surveillance will be conducted after administration of peginterferon alfa-2b (administered according to the directions on the products' labeling). PegIntron Injection for surveillance is a weight-based dosing product administered at a dose of 0.5/1.0 ug/kg or 1.5 ug/kg. Administration of treatment is not part of this study.
  Other Names: PegIntron

SUMMARY:
Surveillance will be conducted at digestive departments of internal medicine in university or general hospitals where participants with chronic hepatitis C are generally treated. The purpose of this surveillance is to evaluate the postmarketing safety and efficacy of PegIntron Injection under actual conditions of use and to examine adverse events, serious adverse events, and adverse drug reactions.

DETAILED DESCRIPTION:
The investigator will record continuously from the first patient since the day of contract to the numbers of patients of contract based on Pegintron approval.

ELIGIBILITY:
Inclusion Criteria:

* Participants with chronic hepatitis C treated with peginterferon alfa-2b.

Signed written contract.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Surveillance will be conducted at digestive departments of internal medicine in university or general hospitals where participants with chronic hepatitis C are generally treated.
Sampling Method: Probability Sample
Enrollment: 1267 (Actual)
Dates: Start 2006-06; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Pegintron/Pegintron Redipen Injection: Participants who have been diagnosed with chronic hepatitis C and treated with PegIntron according to local label.
Period: Overall Study
Arm/Group | Pegintron/Pegintron Redipen Injection
Started | 1267
Completed | 1267
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pegintron/Pegintron Redipen Injection
Number analyzed (Participants) | 1267
Age, Customized [Number; unit: participants]
  Between 16 and 80 years | 1267
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 585
  Male | 682

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Reported a Serious Adverse Event
Description: Serious adverse events (SAE's) were events that resulted in death, were life threatening, required hospitalization, caused disability, and congenital anomaly. All SAE's related or unrelated to the study drug and those SAE's that were determined by the investigator, using specific criteria defined in the protocol, were reported.
Time Frame: 24 weeks after administration of PegIntron Injection
Measure: Number; unit: Participants
Arm/Group | Pegintron/Pegintron Redipen Injection
Number analyzed (Participants) | 1267
Participants | 15

2. Primary Outcome: Number of Participants That Reported a Non Serious Adverse Event Above 5 Percent Threshold
Description: Adverse events (AE's) were events that resulted in unintended signs, symptoms or illnesses. All non-serious adverse events related or unrelated to the study drug and those AE's determined by the investigator, using specific criteria defined in the protocol, were reported.
Time Frame: 24 weeks after administration of PegIntron Injection.
Measure: Number; unit: Participants
Arm/Group | Pegintron/Pegintron Redipen Injection
Number analyzed (Participants) | 1267
Participants | 820

ADVERSE EVENTS:
Arm/Group | Pegintron/Pegintron Redipen Injection
Serious Adverse Events (participants affected / at risk) | 15/1267
Other Adverse Events (participants affected / at risk) | 820/1267
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pegintron/Pegintron Redipen Injection (N=1267)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Cardiac Failure (Cardiac disorders) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Chest Pain (General disorders) | 1 (1)
Bronchiectasis (Infections and infestations) | 1 (1)
Empyema (Infections and infestations) | 1 (1)
Herpes Zoster (Infections and infestations) | 1 (1)
Meningitis Cryptococcal (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Blood Amylase Increased (Investigations) | 1 (1)
Lipase Increased (Investigations) | 1 (1)
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 1 (1)
Hepatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hepatic Neoplasm Malignant Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Coma (Nervous system disorders) | 1 (1)
Homicidal Ideation (Psychiatric disorders) | 1 (1)
Suicide Attempt (Psychiatric disorders) | 1 (1)
Alveolitis Allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pegintron/Pegintron Redipen Injection (N=1267)
Anaemia (Blood and lymphatic system disorders) | 237 (243)
Leukopenia (Blood and lymphatic system disorders) | 144 (152)
Thrombocytopenia (Blood and lymphatic system disorders) | 81 (84)
Dyspepsia (Gastrointestinal disorders) | 102 (112)
Nausea (Gastrointestinal disorders) | 69 (76)
Asthenia (General disorders) | 80 (87)
Fatigue (General disorders) | 70 (76)
Pyrexia (General disorders) | 71 (86)
White Blood Cell Count Decreased (Investigations) | 97 (107)
Decreased Appetite (Metabolism and nutrition disorders) | 124 (137)
Myalgia (Musculoskeletal and connective tissue disorders) | 227 (275)
Headache (Nervous system disorders) | 226 (288)
Insomnia (Psychiatric disorders) | 82 (87)
Alopecia (Skin and subcutaneous tissue disorders) | 82 (84)
Pruritus (Skin and subcutaneous tissue disorders) | 182 (198)
Rash (Skin and subcutaneous tissue disorders) | 70 (77)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No